CLINICAL TRIAL: NCT02604888
Title: Efficacy Study of a Cosmetic Lotion in the Treatment of Alopecia Areata in Males and Females
Acronym: MEXISAREATA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mexis George (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MEXIS-ALOPECIA AREATA-2015
Record Dates: First submitted 2015-11-09; First posted 2015-11-16 (Estimated); Last update posted 2017-01-04 (Estimated); Status verified 2017-01

CONDITIONS: Alopecia Areata
Keywords: Baldness; Alopecia Areata; Alopecia; Hair loss
MeSH Terms: conditions — Alopecia Areata; Alopecia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Volunteers (Other): 20 volunteers both men and women with an age between 18 and 70 years suffering from Alopecia Areata in several types apply on the scalp drops of the MEXIS/M6S PATENT - lotion against Alopecia
  Interventions: Other: MEXIS/M6S Patent - lotion against alopecia

INTERVENTIONS:
Other: MEXIS/M6S Patent - lotion against alopecia — For greatest problems 20 drops on the scalp per day for 6 months. For minor problems 10 drops on the scalp three times per week for 6 months.

SUMMARY:
The purpose of this study is to determine whether the Hair Loss Prevention Lotion named MEXIS, M.P.A.F., M6S PATENT is effective in the treatment of Alopecia Areata.

DETAILED DESCRIPTION:
This study verifies whether the tested product has any efficacy in the treatment of Alopecia Areata.

* The evaluated product (Hair Loss prevention Lotion) is called: MEXIS, MPAF, M6S PATENT.
* 20 volunteers both men and women suffering from hair loss both in parties and over the entire scalp with age between 18 and 70 years will be selected for this test .
* Samples of the product have been applied following their usual use: as they are.
* On the selecting volunteers will be used:

A polarized light video-camera to check the redness of the scalp and to have a picture of hair and scalp.

* Volunteers will also be asked about:
* Fluffiness
* Sheen
* Itching
* Presence of scales on scalp
* Oily hair
* Product's acceptability
* The readings will be taken at 0 time (basal value), after 15 days (t15), 30 days (t30), 45 days (t45), 45 days (t45), 60 days (t60) and 90 days (t90) by the experimenter in the medical studio. Then they analyzed and reported in a graph.
* Summarizing tables and graphs of the data will be taken during experimentation.

ELIGIBILITY:
Inclusion Criteria:

* Good state of general health
* Suffering from Alopecia Areata
* No pharmacological treatment in progress
* Promise not to change the usual daily routine
* No atopy in the anamnesis

Exclusion Criteria:

* Illness
* Good state of hair
* Pharmacological treatment in progress
* Denial of the continuance of the usual daily routine
* Atopy in the anamnesis

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2015-10; Primary Completion 2016-10 (Actual); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
Change of the Density of the Hair measured with a camera | baseline and 180 days
  Change on the total amount of head's hair

SECONDARY OUTCOMES:
Change of the Amount of Hair Loss | baseline and 180 days
  Change on the amount of hair fallen per day

CONTACTS AND LOCATIONS:
Overall Officials: Markos Papakonstantis, Monitor, Study Chair — 401 General Military Hospital of Athens, Dermatology clinic
Locations (1):
- George Mexis, Athens, Greece

IPD SHARING:
Plan to Share IPD: Yes